CLINICAL TRIAL: NCT01771224
Title: Effect of Palmitoleic Acid (FAn-7) on Expression of HNF4γ and Ulcerative Colitis (UC) Activity
Brief Title: Effect of FAn-7 in UC Activity
Acronym: FAUC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Jesús Kazuo Yamamoto Furusho, MD PhD, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REF453
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: Palmitoleic acid ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — palmitoleic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- palmitoleic acid (Experimental): Palmitoleic acid: 720 mg/day for 56 days
  Interventions: Dietary Supplement: Palmitoleic acid
- Sugar pill (Placebo Comparator): Sugar pill: 720 mg/day for 56 days

INTERVENTIONS:
Dietary Supplement: Palmitoleic acid — Palmitoleic acid and 5-ASA
  Arms: palmitoleic acid

SUMMARY:
Introduction: Inflammatory bowel disease (IBD) refers to two chronic diseases that cause intestinal inflammation, ulcerative colitis (UC) and Crohn's disease (CD). The conventional treatment is not effective; therefore, alternative therapies may be effective specially in UC patients. Fatty acid (FA) may have a beneficial effect on some UC patients. The increasing incidence and prevalence of UC and ineffective treatments in some patients, allows search coadjuvant therapies. Objective: Quantification of differences between patients with and without FA. Methods: In two groups of patients with UC is administered FA and placebo. We will measure the changes clinical, endoscopic and histological in both groups, before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histopathologically confirmed diagnosis of UC.
* With mild and moderate disease.
* Patients treated with only doses of 5-aminosalicylates (5-ASA)
* BMI, 18 to 34.9 kg/m2
* Born in Mexico the last two generations
* Each patient will be asked to sign and date the consent form, to indicate that you agree to participate.

Exclusion Criteria:

* Patient with associated diseases such as diabetes mellitus, hypertension, dyslipidemia, atherosclerosis and malabsorption syndrome.
* With autoimmune diseases (lupus, HIV, cancer and hepatitis), colitis (infectious, post-radiation, post-drug, indeterminate) and Crohn's Disease.
* If the patient use drugs that inhibit fat absorption.
* Patients after partial or total resection of stomach or small intestine.
* Steroid users.
* Patients in remission histology, clinical and endoscopic.
* Patients treated with FAn-3,6 or 9.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
clinical and endoscopic remission | 2 months
  We will perfom a basal and final colonoscopy

SECONDARY OUTCOMES:
quantification IL-6 in colonic mucosa | 2 months
  quantification of IL-6 by RT-PCR in colonic mucosa at before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús K Yamamoto, MD, PhD, Study Director — Inflammatory Bowel Disease Clinic; Nallely Bueno, MSc, Principal Investigator — Inflammatory Bowel Disease Clinic
Locations (1):
- INCMNSZ, DF, Tlalpan, Mexico

REFERENCES:
- [Result] Bueno-Hernandez N, Sanchez-Munoz F, Barreto-Zuniga R, Dominguez-Lopez A, Yamamoto-Furusho JK. Expression of HNF4gamma is downregulated in patients with active ulcerative colitis (UC) compared to UC patients in remission and healthy controls. Inflamm Bowel Dis. 2011 Aug;17(8):E91. doi: 10.1002/ibd.21753. Epub 2011 May 25. No abstract available. PMID 21618351
- [Result] Drewes T, Senkel S, Holewa B, Ryffel GU. Human hepatocyte nuclear factor 4 isoforms are encoded by distinct and differentially expressed genes. Mol Cell Biol. 1996 Mar;16(3):925-31. doi: 10.1128/MCB.16.3.925. PMID 8622695
- [Result] Gruber L, Lichti P, Rath E, Haller D. Nutrigenomics and nutrigenetics in inflammatory bowel diseases. J Clin Gastroenterol. 2012 Oct;46(9):735-47. doi: 10.1097/MCG.0b013e31825ca21a. PMID 22941427
- [Result] Daigo K, Kawamura T, Ohta Y, Ohashi R, Katayose S, Tanaka T, Aburatani H, Naito M, Kodama T, Ihara S, Hamakubo T. Proteomic analysis of native hepatocyte nuclear factor-4alpha (HNF4alpha) isoforms, phosphorylation status, and interactive cofactors. J Biol Chem. 2011 Jan 7;286(1):674-86. doi: 10.1074/jbc.M110.154732. Epub 2010 Nov 3. PMID 21047794
- [Result] Nieto N, Torres MI, Rios A, Gil A. Dietary polyunsaturated fatty acids improve histological and biochemical alterations in rats with experimental ulcerative colitis. J Nutr. 2002 Jan;132(1):11-9. doi: 10.1093/jn/132.1.11. PMID 11773501
- [Result] Nishida T, Miwa H, Shigematsu A, Yamamoto M, Iida M, Fujishima M. Increased arachidonic acid composition of phospholipids in colonic mucosa from patients with active ulcerative colitis. Gut. 1987 Aug;28(8):1002-7. doi: 10.1136/gut.28.8.1002. PMID 3117625
- [Result] Ahn SH, Shah YM, Inoue J, Morimura K, Kim I, Yim S, Lambert G, Kurotani R, Nagashima K, Gonzalez FJ, Inoue Y. Hepatocyte nuclear factor 4alpha in the intestinal epithelial cells protects against inflammatory bowel disease. Inflamm Bowel Dis. 2008 Jul;14(7):908-20. doi: 10.1002/ibd.20413. PMID 18338782
- [Result] Taraviras S, Mantamadiotis T, Dong-Si T, Mincheva A, Lichter P, Drewes T, Ryffel GU, Monaghan AP, Schutz G. Primary structure, chromosomal mapping, expression and transcriptional activity of murine hepatocyte nuclear factor 4gamma. Biochim Biophys Acta. 2000 Jan 31;1490(1-2):21-32. doi: 10.1016/s0167-4781(99)00232-8. PMID 10786614
- [Result] Watanabe T, Kobunai T, Toda E, Kanazawa T, Kazama Y, Tanaka J, Tanaka T, Yamamoto Y, Hata K, Kojima T, Yokoyama T, Konishi T, Okayama Y, Sugimoto Y, Oka T, Sasaki S, Ajioka Y, Muto T, Nagawa H. Gene expression signature and the prediction of ulcerative colitis-associated colorectal cancer by DNA microarray. Clin Cancer Res. 2007 Jan 15;13(2 Pt 1):415-20. doi: 10.1158/1078-0432.CCR-06-0753. PMID 17255260
- [Result] Wille JJ, Kydonieus A. Palmitoleic acid isomer (C16:1delta6) in human skin sebum is effective against gram-positive bacteria. Skin Pharmacol Appl Skin Physiol. 2003 May-Jun;16(3):176-87. doi: 10.1159/000069757. PMID 12677098
- [Result] Wisely GB, Miller AB, Davis RG, Thornquest AD Jr, Johnson R, Spitzer T, Sefler A, Shearer B, Moore JT, Miller AB, Willson TM, Williams SP. Hepatocyte nuclear factor 4 is a transcription factor that constitutively binds fatty acids. Structure. 2002 Sep;10(9):1225-34. doi: 10.1016/s0969-2126(02)00829-8. PMID 12220494
- [Result] Okuma Y, Shirao T, Sakamoto A. [Constipation in intracranial diseases--correlation betweeen the cerebrospinal fluid pressure and constipation]. Saishin Igaku. 1971 Jan;26(1):139-44. No abstract available. Japanese. PMID 5539258
- [Result] Wu F, Dassopoulos T, Cope L, Maitra A, Brant SR, Harris ML, Bayless TM, Parmigiani G, Chakravarti S. Genome-wide gene expression differences in Crohn's disease and ulcerative colitis from endoscopic pinch biopsies: insights into distinctive pathogenesis. Inflamm Bowel Dis. 2007 Jul;13(7):807-21. doi: 10.1002/ibd.20110. PMID 17262812